CLINICAL TRIAL: NCT06698497
Title: Boosting COVID-19 Vaccination Uptake Using Wastewater Surveillance: A County-Randomized Controlled Trial
Brief Title: Boosting COVID-19 Vaccination Uptake Using Wastewater Surveillance
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Syracuse University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: 23-327
Record Dates: First submitted 2024-11-08; First posted 2024-11-21 (Actual); Last update posted 2025-09-15 (Actual); Status verified 2025-09

CONDITIONS: Vaccine Uptake
Keywords: COVID-19 vaccine; wastewater surveillance; vaccine campaign; communication campaign; vaccine uptake; vaccine hesitancy; health belief model; COVID-19; SARS-CoV-2; coronavirus
MeSH Terms: conditions — Vaccination Hesitancy; COVID-19; Coronavirus Infections

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Communications Intervention Group (Experimental)
  Interventions: Behavioral: Communication Campaign
- Control (No Intervention)

INTERVENTIONS:
Behavioral: Communication Campaign — A social media vaccine communications campaign is deployed once increasing amounts of SARS-CoV-2 RNA are identified in the New York State wastewater surveillance network. The social media campaigns on Facebook, Instagram, and NextDoor social media platforms will run for 11 weeks. The campaign disseminates information about the wastewater surveillance network and vaccination (not COVID-19 specific) to residents in intervention counties. These social media platforms not only allow for quick and cost-effective exposure, but also allow for participation and interaction with participants. The campaign ads include a call-to-action link to the New York State wastewater surveillance network webpage which has information and links regarding vaccines for respiratory transmitted pathogens (COVID-19, influenza, and RSV) and how to schedule an appointment.
  Arms: Communications Intervention Group

SUMMARY:
Vaccinations are among the most successful and critical public health interventions. Despite the enormous protection that vaccines provide to public health, both delays and refusals of vaccines (vaccine hesitancy) are on the rise. Given that low vaccination rates present both an individual and community risk, it is critical that measures are taken to increase vaccination uptake in both rural and urban counties in New York. Wastewater surveillance of SARS-CoV-2 has been shown to be a leading indicator of pending surges. This study will examine whether a communications campaign based upon SARS-CoV-2 wastewater surveillance data can increase COVID-19 vaccine uptake.

Forty counties have been selected for the communication campaign (20 in the treatment group and 20 in the control group). A difference-in-differences method will be applied to assess the impact of the communications campaign on vaccine uptake, which observes the outcomes between a control and treatment group over pre- and post-intervention time periods. The communications campaign will be evaluated using the change in vaccination status of residents of the treatment and control counties. Outcomes will also be compared between demographic groups including race and ethnicity because of differences in vaccination rates that have been already observed.

We hypothesize that information regarding COVID-19 provided by wastewater surveillance that is geographically based and more local to communities will increase COVID-19 vaccine uptake. This theory of local information having an impact on health behavior is a novel application of the health belief model to increase vaccine uptake.

ELIGIBILITY:
Inclusion Criteria:

* Counties in New York State

Exclusion Criteria:

* Counties outside of New York State

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2024-09-13 (Actual); Primary Completion 2024-11-24 (Actual); Study Completion 2025-07-10 (Actual)

PRIMARY OUTCOMES:
COVID-19 Vaccine Uptake | 11 weeks
  The change in vaccination coverage among residents of the counties in the study will be measured as the percent of the population that received a vaccine dose.

CONTACTS AND LOCATIONS:
Locations (1):
- Syracuse University, Syracuse, New York, United States